CLINICAL TRIAL: NCT05112419
Title: A Single Dose, Non-Randomised, Open-Label, Parallel-Group Study to Investigate the Pharmacokinetics, Safety, and Tolerability of Zibotentan in Healthy Participants Compared to Participants With Moderate Hepatic and Moderate Renal Impairment
Brief Title: A Study to Assess Zibotentan Pharmacokinetics in Participants With Moderate Hepatic and Moderate Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4326C00001; 2021-003289-10 (EudraCT Number)
Record Dates: First submitted 2021-10-11; First posted 2021-11-08 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hepatic Impairment; Renal Impairment
Keywords: Renal Impairment; Hepatic Impairment; Healthy participants; Zibotentan; Pharmacokinetics; Safety
MeSH Terms: conditions — Renal Insufficiency | interventions — ZD4054

STUDY DESIGN:
Intervention Model Description: Two cohorts (patients and matched healthy subjects) to be enrolled for this study.
  Approximately 12 participants will be enrolled into each one of the 2 cohorts and receive the study intervention:
  * Cohort 1 will enroll participants with moderate hepatic impairment and moderate renal impairment as assessed at screening.
  * Cohort 2 will enroll healthy participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Participants with moderate hepatic impairment and moderate renal impairment (Experimental): Participants will receive a single oral dose of zibotentan under fasted conditions.
  Interventions: Drug: Zibotentan
- Cohort 2: Healthy participants (Experimental): Participants will receive a single oral dose of zibotentan under fasted conditions.
  Interventions: Drug: Zibotentan

INTERVENTIONS:
Drug: Zibotentan — All participants will receive a single oral dose of zibotentan capsule under fasted conditions.

SUMMARY:
This study will evaluate the pharmacokinetics (PK), safety, and tolerability of a single oral dose of zibotentan in patients with moderate hepatic and moderate renal impairment in comparison to a matched healthy control group.

DETAILED DESCRIPTION:
This is a single-dose, non-randomised, open-label, parallel-group study.

All participants will receive a single oral dose of 5 mg zibotentan under fasted conditions and will be involved in the study for approximately 5 weeks.

Approximately 12 participants will be enrolled into each one of the 2 cohorts and receive the study intervention:

* Cohort 1: 12 participants with moderate hepatic impairment and moderate renal impairment as assessed at Screening
* Cohort 2: 12 healthy participants matched for age (± 10 years), gender, and BMI (± 20%) on a group level to participants in Cohort 1

The study will comprise of the following study periods:

* A Screening Period of maximum 28 days (before dosing): participants will be screened for eligibility.
* A Residential Period of 8 days: participants will be admitted to the study centre in the evening on Day
* 2, two days before administration of a single oral dose of zibotentan (Day 1). Participants will have final study assessments on Day 6 (120 hours post-dose) and will be discharged that day.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of at least 50 kg and body mass index within the range of 18 and 35 kg/m^2 (inclusive).
* Female of non-childbearing potential or male

Participants with Moderate Hepatic Impairment and Moderate Renal Impairment only (Cohort 1)

* An estimated glomerular filtration rate (eGFR) in the range of 30 to 45 mL/min/1.73m^2 (inclusive) as determined using the Chronic Kidney Disease Epidemiology Collaboration formula, at Screening. Retesting for eGFR may be repeated twice during Screening Period.
* Confirmed clinical diagnosis of cirrhosis with either ascites or moderate hepatic impairment (Childs-Pugh B). Supporting documents confirming the participant's hepatic impairment must be available. The participant must be classified by the Investigator or usual practitioner as Child-Pugh Class B or having radiographic or clinical evidence of ascites of any grade.
* Stable hepatic impairment (eg, no clinically significant change in signs, symptoms, or laboratory parameters of hepatic disease status within 28 days prior to Screening, as determined by the Investigator or usual practitioner).

Healthy Participants only (Cohort 2)

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and clinical laboratory tests.
* An eGFR of ≥ 90 mL/min/1.73m^2 as determined using the CKD-EPI formula at Screening.
* No clinically significant liver or kidney disease as judged by the Investigator.

Exclusion Criteria:

Medical Conditions

* Any evidence of a clinically significant disease which in the Investigator's opinion makes it undesirable for the participant to participate in the study.
* History of alcohol abuse or excessive intake of alcohol within 6 months prior to the Screening visit. Definition of excessive intake: an average weekly intake of >7 drinks/week for men or > 3.5 drinks/week for women. One drink is equivalent to (16 g of alcohol).
* Positive alcohol or drug of abuse at Screening.
* Participants with a history of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator, to drugs with a similar chemical structure or class to zibotentan.
* Participants with known hypersensitivity/allergic reaction to paracetamol.
* Any signs or confirmation of coronavirus disease-19 infection.

Participants with Moderate Hepatic Impairment and Moderate Renal Impairment only (Cohort 1)

* Presence of unstable medical (eg, diabetes, epilepsy) or psychological conditions which, in the opinion of the Investigator, would compromise the participant's safety or successful participation in this study.
* Fluctuating or rapidly deteriorating hepatic function, as indicated by strongly varying or worsening of clinical and/or laboratory signs of hepatic impairment within 28 days prior to dosing (eg, infection of ascites, fever, or active gastrointestinal bleeding).
* Severe hepatic impairment (Child-Pugh Class C Hepatic impairment), an isolated aspartate aminotransferase (AST) or alanine aminotransferase (ALT)> 5 x the upper limit of normal (ULN); or total bilirubin > 2 x ULN at time of enrolment or a concurrent increased AST and ALT of > 3 x the ULN together with a total bilirubin of > 2 x ULN. An isolated increase in bilirubin in participants with known Gilbert's syndrome is not a reason for exclusion.
* Acute liver disease caused by drug toxicity or by an infection.
* Presence of a hepatocellular carcinoma.
* Liver or renal transplantation or planned within the next 3 months at Screening.
* Receiving renal replacement therapy.
* Recent acute or subacute renal function deterioration (eg, participants with large fluctuations of creatinine values, as judged by the Investigator, and documented within 28 days prior to Screening).
* New York Heart Association functional heart failure Class III or intravenous or with unstable heart failure requiring hospitalisation for optimisation of heart failure treatment and who are not yet stable on heart failure therapy within 6 months prior to Screening.
* Abnormal resting vital signs (after resting for 10 minutes) of supine systolic blood pressure> 180 mmHg or < 100 Hg; or diastolic blood pressure> 110 mmHg or < 50 mmHg.
* Change in dose regimen of medically-required medication within the 14 days before dosing.

Healthy Participants only (Cohort 2)

- History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.

Prior/Concomitant Therapy

* Use of strong or moderate inhibitors or inducers of CYP3A4 within 28 days prior to dose of zibotentan.
* Use of phosphate binders (eg, aluminium hydroxide and calcium carbonate) and acid reducing agents such as cholestyramine/colestipol, ranitidine/nizatidine, or proton pump inhibitors within 3 days before and 12 hours after dosing with zibotentan.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Area under plasma concentration-time curve from time zero to infinity (AUCinf) | Day 1 to Day 6
  To assess the PK of a single oral dose of zibotentan in participants with moderate hepatic impairment and moderate renal impairment compared to a group of healthy matched controls
Area under the plasma concentration-curve from time zero to time of last quantifiable concentration (AUClast) | Day 1 to Day 6
  To assess the PK of a single oral dose of zibotentan in participants with moderate hepatic impairment and moderate renal impairment compared to a group of healthy matched controls
Maximum observed plasma concentration (Cmax) | Day 1 to Day 6
  To assess the PK of a single oral dose of zibotentan in participants with moderate hepatic impairment and moderate renal impairment compared to a group of healthy matched controls

SECONDARY OUTCOMES:
Number of participants with adverse events | Screening (Day -28 to Day -2) to Day 6
  To evaluate the safety and tolerability of a single oral dose of zibotentan in participants with moderate hepatic impairment and moderate renal impairment compared to a group of healthy matched controls
Time to reach maximum observed plasma concentration (tmax) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Area under the plasma concentration-time curve from time zero to 24 hours post-dose (AUC[0-24]) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Area under plasma concentration-time curve from time zero to 72 hours post-dose (AUC [0-72]) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Half-life associated with terminal slope (λz) of a semi-logarithmic concentration-time curve (t½λz) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Terminal elimination rate constant (λz) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Apparent total body clearance of drug from plasma after extravascular administration (CL/F) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Apparent total non-renal body clearance of drug from plasma after extravascular administration (CLNR/F) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) | Day 1 to Day 6
  To further characterise zibotentan plasma PK in all treatment groups
Amount of unchanged drug excreted into urine from time t1 to time t2 [Ae (t1-t2)] | Day 1 to Day 3
  To further characterise zibotentan urine PK in all treatment groups
Cumulative amount of unchanged drug excreted into urine from time of dosing (time 0) through time t [Ae (0-t)] | Day 1 to Day 3
  To further characterise zibotentan urine PK in all treatment groups
Percentage of dose excreted unchanged in urine from time t1 to time t2 [fe (t1-t2)] | Day 1 to Day 3
  To further characterise zibotentan urine PK in all treatment groups
Percentage of dose excreted unchanged in urine from time of dosing (time 0) through time t [fe (0-t)] | Day 1 to Day 3
  To further characterise zibotentan urine PK in all treatment groups
Renal clearance of drug from plasma, calculated as Ae0-t/AUC0-t where t is matched for urine and plasma (CLR) | Day 1 to Day 3
  To further characterise zibotentan urine PK in all treatment groups

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Mercier AK, Sunnaker M, Ueckert S, Pawlik T, Henricson E, Molodetskyi O, Law GC, Parker VER, Oscarsson J. Pharmacokinetics and Tolerability of Zibotentan in Patients with Concurrent Moderate Renal and Moderate Hepatic Impairment. Clin Pharmacokinet. 2023 Dec;62(12):1713-1724. doi: 10.1007/s40262-023-01306-7. Epub 2023 Oct 6. PMID 37801266